CLINICAL TRIAL: NCT06739486
Title: Efficacy of Sodium Glucose Cotransporter 2 Inhibitors on Non-Alcoholic Fatty Liver Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdallah Gamal Eldin Shawky Mohamed Hamad, Internal resident, Assiut University
Other Study IDs: SGLT.2 inhibitors
Record Dates: First submitted 2024-11-17; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Non Alcholic Fatty Liver Disease; Hepatic Steatosis; Hepatic Fibrosis; NAFLD (Nonalcoholic Fatty Liver Disease)
Keywords: NAFLD; Non alcoholic fatty liver disease; Hepatic steatosis; Hepatic fibrosis; Na glucose cotransporter 2 inhibitors; SGLT-2 inhibitors
MeSH Terms: conditions — Fatty Liver; Liver Cirrhosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
evaluate the effectiveness of sodium-glucose cotransporter-2 (SGLT.2) inhibitors in improving hepatic steatosis and hepatic fibrosis using imaging biomarkers and histopathology in patients with non-alcoholic fatty liver disease

DETAILED DESCRIPTION:
2.1 Background (Research Question, Available Data from the literature, Current strategy for dealing with the problem, Rationale of the research that paves the way to the aim(s) of the work). (200-250 words max.) Non-alcoholic fatty liver disease (NAFLD) is a leading cause of liver-related health issues worldwide, with prevalence rates reaching up to 30%.The number of cases has been steadily rising, increasing from 391.2 million in 1990 to 882.1 million in 2017.

NAFLD is often linked to one or more components of metabolic syndrome, such as hypertension, dyslipidemia, obesity, and Type 2 diabetes mellitus, along with insulin resistance. Although the exact pathogenesis of NAFLD is not fully understood, there is increasing evidence that insulin resistance and lipid metabolism dysregulation play significant roles in the development of hepatic steatosis. Factors such as a high-fat diet, insulin resistance, obesity, and dysregulated peripheral lipolysis contribute to the increased influx of free fatty acids into the liver, leading to a 'lipotoxic' state within hepatocytes.The accumulation of triacylglycerol in the cytoplasm of hepatocytes manifests histologically as steatosis. Persistent micro-hepatic injury eventually results in endoplasmic reticulum stress and mitochondrial dysfunction, which then contribute to lobular inflammation, cellular apoptosis, and hepatic fibrosis over time.

If left untreated, this manageable condition can lead to serious complications, including advanced cirrhosis, hepatocellular carcinoma, and potentially cardiovascular morbidity.and mortality.Given the serious prognostic implications of NAFLD, effective treatment is essential to prevent disease progression. While weight loss and lifestyle modifications are the primary treatments, pharmacologic options remain limited. Recently, the potential of a novel oral hypoglycemic agent known as sodium-glucose cotransporter 2 (SGLT-2) inhibitors in the treatment of NAFLD has been explored through various animal studies on rodent models and human clinical trials, showing promising effects.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* both sex

Exclusion Criteria:

* alcohol drinker
* any cause of liver affection (hepatitis, autoimmune…etc)
* patients with kidney function affection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged over 18 years, not alcohol drinker,has any cause of liver affection,or with kidney function affection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
determine the effects of dapagliflozin, an SGLT2 inhibitor, on hepatic fibrosis and steatosis in patients with NAFLD using fibroscan and biomarkers | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah A Gamal, Resident, Principal Investigator — Assiut University; Lobna A Farag, Lecturer, Study Director — Assiut University; Mohamed A Abozaid, Lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Foucher J, Chanteloup E, Vergniol J, Castera L, Le Bail B, Adhoute X, Bertet J, Couzigou P, de Ledinghen V. Diagnosis of cirrhosis by transient elastography (FibroScan): a prospective study. Gut. 2006 Mar;55(3):403-8. doi: 10.1136/gut.2005.069153. Epub 2005 Jul 14. PMID 16020491
- [Background] Ge X, Zheng L, Wang M, Du Y, Jiang J. Prevalence trends in non-alcoholic fatty liver disease at the global, regional and national levels, 1990-2017: a population-based observational study. BMJ Open. 2020 Aug 3;10(8):e036663. doi: 10.1136/bmjopen-2019-036663. PMID 32747349
- [Background] Younossi ZM, Golabi P, de Avila L, Paik JM, Srishord M, Fukui N, Qiu Y, Burns L, Afendy A, Nader F. The global epidemiology of NAFLD and NASH in patients with type 2 diabetes: A systematic review and meta-analysis. J Hepatol. 2019 Oct;71(4):793-801. doi: 10.1016/j.jhep.2019.06.021. Epub 2019 Jul 4. PMID 31279902
- [Background] Li X, Wang H. Multiple organs involved in the pathogenesis of non-alcoholic fatty liver disease. Cell Biosci. 2020 Dec 7;10(1):140. doi: 10.1186/s13578-020-00507-y. PMID 33372630
- [Background] Adams LA, Lymp JF, St Sauver J, Sanderson SO, Lindor KD, Feldstein A, Angulo P. The natural history of nonalcoholic fatty liver disease: a population-based cohort study. Gastroenterology. 2005 Jul;129(1):113-21. doi: 10.1053/j.gastro.2005.04.014. PMID 16012941
- [Background] Soderberg C, Stal P, Askling J, Glaumann H, Lindberg G, Marmur J, Hultcrantz R. Decreased survival of subjects with elevated liver function tests during a 28-year follow-up. Hepatology. 2010 Feb;51(2):595-602. doi: 10.1002/hep.23314. PMID 20014114
- [Background] Tahara A, Takasu T. SGLT2 inhibitor ipragliflozin alone and combined with pioglitazone prevents progression of nonalcoholic steatohepatitis in a type 2 diabetes rodent model. Physiol Rep. 2019 Nov;7(22):e14286. doi: 10.14814/phy2.14286. PMID 31782258
- [Background] Wei Q, Xu X, Guo L, Li J, Li L. Effect of SGLT2 Inhibitors on Type 2 Diabetes Mellitus With Non-Alcoholic Fatty Liver Disease: A Meta-Analysis of Randomized Controlled Trials. Front Endocrinol (Lausanne). 2021 Jun 17;12:635556. doi: 10.3389/fendo.2021.635556. eCollection 2021. PMID 34220701
- [Background] Jojima T, Tomotsune T, Iijima T, Akimoto K, Suzuki K, Aso Y. Empagliflozin (an SGLT2 inhibitor), alone or in combination with linagliptin (a DPP-4 inhibitor), prevents steatohepatitis in a novel mouse model of non-alcoholic steatohepatitis and diabetes. Diabetol Metab Syndr. 2016 Jul 26;8:45. doi: 10.1186/s13098-016-0169-x. eCollection 2016. PMID 27462372
- [Background] Arai T, Atsukawa M, Tsubota A, Mikami S, Ono H, Kawano T, Yoshida Y, Tanabe T, Okubo T, Hayama K, Nakagawa-Iwashita A, Itokawa N, Kondo C, Kaneko K, Emoto N, Nagao M, Inagaki K, Fukuda I, Sugihara H, Iwakiri K. Effect of sodium-glucose cotransporter 2 inhibitor in patients with non-alcoholic fatty liver disease and type 2 diabetes mellitus: a propensity score-matched analysis of real-world data. Ther Adv Endocrinol Metab. 2021 Mar 21;12:20420188211000243. doi: 10.1177/20420188211000243. eCollection 2021. PMID 33815743
- [Background] Shimizu M, Suzuki K, Kato K, Jojima T, Iijima T, Murohisa T, Iijima M, Takekawa H, Usui I, Hiraishi H, Aso Y. Evaluation of the effects of dapagliflozin, a sodium-glucose co-transporter-2 inhibitor, on hepatic steatosis and fibrosis using transient elastography in patients with type 2 diabetes and non-alcoholic fatty liver disease. Diabetes Obes Metab. 2019 Feb;21(2):285-292. doi: 10.1111/dom.13520. Epub 2018 Oct 2. PMID 30178600
- [Background] Adams LA, Anstee QM, Tilg H, Targher G. Non-alcoholic fatty liver disease and its relationship with cardiovascular disease and other extrahepatic diseases. Gut. 2017 Jun;66(6):1138-1153. doi: 10.1136/gutjnl-2017-313884. Epub 2017 Mar 17. PMID 28314735
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365